CLINICAL TRIAL: NCT01613287
Title: A Clinical Proof of Concept Study of IMMUNOadsorption Therapy in Patients With Idiopathic Pulmonary Arterial Hypertension
Brief Title: Proof of Concept Study of IMMUNOadsorption Therapy in Patients With Idiopathic Pulmonary Arterial Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Miltenyi Biotec B.V. & Co. KG (Industry)
Responsible Party: Sponsor
Organization: Miltenyi Biomedicine GmbH (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M-2010-224; CIV-11-10-002861 (Other: European Databank on Medical Devices - EUDAMED)
Record Dates: First submitted 2012-05-29; First posted 2012-06-07 (Estimated); Last update posted 2020-07-10 (Actual); Status verified 2013-12

CONDITIONS: Idiopathic Pulmonary Arterial Hypertension
Keywords: Pulmonary Hypertension; Pulmonary Arterial Hypertension; TheraSorb; immunoadsorption
MeSH Terms: conditions — Familial Primary Pulmonary Hypertension; Hypertension, Pulmonary; Pulmonary Arterial Hypertension | interventions — Plasmapheresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Immunoadsorption (Experimental): Patients are treated with the TheraSorb® Ig flex adsorber used exclusively with the LIFE 18® apheresis system for extracorporeal application for IA therapy (5 treatments) performed over 5 to 8 consecutive days
  Interventions: Device: TheraSorb® - Ig flex

INTERVENTIONS:
Device: TheraSorb® - Ig flex — TheraSorb® Treatment with one TheraSorb® Ig flex adsorber pair, used exclusively with the LIFE 18® apheresis system for extracorporeal application for IA therapy.
  5 treatments performed over 5 to 8 consecutive days.
  Other Names: Immunoadsorption

SUMMARY:
This clinical investigation is a medical device trial to examine the safety and efficacy of TheraSorb® Ig flex adsorber treatment (as an add-on to conventional treatment) used exclusively with the LIFE 18® apheresis system for extracorporeal application for IA therapy (5 treatments) performed over 5 to 8 consecutive days in patients with Idiopathic Pulmonary Arterial Hypertension and WHO functional classification III.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and willing to sign the Informed Consent Form
* age > 18 and < 80 years at time of informed consent
* Idiopathic pulmonary arterial hypertension diagnosed by right heart catheter
* WHO functional classification III
* Application of conventional IPAH therapy, which has been stable for the prior 8 weeks
* Able to perform a 6-minute-walk test (MWT)
* Negative pregnancy test (β-HCG) at the start of the trial and appropriate contraception throughout the trial for women with child-bearing potential.

Exclusion Criteria:

* Pregnancy and/or lactation
* PAH of any cause other than permitted in the inclusion criteria, e.g. concomitantly to portal hypertension, complex congenital heart disease, reversed shunt, HIV infection, suspected pulmonary veno-occlusive disease
* Contraindication for right heart catheterization
* Any change in disease-targeted therapy within 8 weeks prior to inclusion
* Walking impairment due to causes other than IPAH that would preclude performance of a 6MWT
* Any patient who has received any investigational medication within 8 weeks prior to the start of this trial or who is scheduled to receive another investigational drug during the course of the trial between visits V1 and V9
* Known intolerance to immunoadsorption in general or to one of the excipients (e.g. sheep antibodies or agarose) or other supporting agents
* Hemoglobin concentration of < 75% below the lower limit of normal
* Systolic blood pressure < 85 mmHg
* Lack of compliance or other similar reason that, in the judgment of the Investigator, precludes satisfactory participation in the trial
* Concurrent severe or uncontrolled medical disease (i.e. uncontrolled diabetes, congestive heart failure, myocardial infarction within 6 months prior to the study, unstable and uncontrolled hypertension, chronic renal disease, or active uncontrolled generalized viral, bacterial and/ or mycotic infection) which by assessment of the treating Investigator could compromise patients safety or participation in the study
* Drug or alcohol abuse within the last 5 years
* Hypercoagulability
* Known severe immunodeficiency (e.g. AIDS)
* Severe lung disease: FEV1/FVC < 50%, total capacity < 60% of normal value
* Indications that prohibit transient anticoagulation using Heparin and/or ACD-A-solutions

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-06; Primary Completion 2013-08 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Primary endpoint is the change of pulmonary vascular resistance (PVR) at rest before immunoadsorption compared to 3 months after immunoadsorption therapy determined by right heart catheterization (RHC). | Baseline, 3 months after therapy

SECONDARY OUTCOMES:
all-cause mortality | ~6months
  The patients will be followed for the duration of the study participation, an expected average of 6 months.
occurrence and number of Adverse Events | ~6 months
  The patients will be followed for the duration of the study participation, an expected average of 6 months.
Six-minute walk test (6MWT) | Measurements at baseline, ~1 week, ~1 month, ~3 months and ~6 months after start of therapy
Quality of life questionnaires | Measurements at baseline, and after ~1 month, ~3 months, ~6 months
  SF-36 EQ-5D™
WHO functional classification | Measurements at baseline, ~1 week, ~1 month, ~3 months and ~6 months after start of therapy
  WHO functional classification of pulmonary hypertension (according to the Evian Symposium,1998, modified New York Heart Association (NYHA) Classification
Analysis of Hemodynamics by right heart catheterization: RAP, PAPm, CO, CI, SvO2; sPAP | Measurements at baseline, after ~3 months
  (Right atrial pressure, mean pulmonary arterial pressure, pulmonary capillary wedge pressure, cardiac output, cardiac index, venous oxygen saturation, systolic pulmonary arterial pressure.)
Reduction of IgG | Measurements at baseline, during each treatment visit, ~1 week, ~1 month and ~3 months after start of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ekkehard Grünig, Prof. Dr., Principal Investigator — Heidelberg University
Locations (4):
- Germany (4):
  - Thoraxklinik am Universitätsklinikum Heidelberg in cooperation with Nierenzentrum Heidelberg, Heidelberg, Baden-Wurttemberg
  - Universitätsmedizin Greifswald, Zentrum für Innere Medizin, Klinik und Poliklinik für Innere Medizin B, Greifswald, Mecklenburg-Vorpommern
  - Herzzentrum der Universität zu Köln, Klinik III für Innere Medizin und Zentrum für Molekulare Medizin, Cologne, North Rhine-Westphalia
  - Deutsches Herzzentrum Berlin, Klinik für Herz-, Thorax- und Gefäßchirurgie, Berlin